CLINICAL TRIAL: NCT04746027
Title: Empathy, Psychopathy and Autism: Behavioural Associations and the Role of an Oxytocin Receptor Polymorphism in a Non-clinical Population
Brief Title: Empathy, Psychopathy and Autism: Behavioural Associations and the Role of an Oxytocin Receptor Polymorphism in a Non-clinical Adult Population
Status: Completed | Type: Observational
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2016-17_092
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-01

CONDITIONS: Empathy; Autism; Psychopathy
Keywords: psychology; biopsychology; genetics
MeSH Terms: conditions — Autistic Disorder; Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples extracted from saliva samples. These samples were collected via passive drool.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an investigation into the associations between psychopathic traits, autistic traits and empathy (cognitive and affective) in the general population as measured using three self report questionnaires and one behavioural task. Participants will also be genotyped for OXTR rs53576 to assess whether this mutation associates with any of the behavioural traits investigated.

DETAILED DESCRIPTION:
In clinical populations with psychopathy or autism, associations with different forms of empathy have been found. An increase in autistic traits has been found to be associated with a decrease in cognitive empathy traits but no difference in affective empathy traits, while an increase in psychopathic traits has been found to be associated with a decrease in both cognitive and affective empathy traits. The current investigation is to establish whether this previously observed relationship between cognitive empathy, affective empathy, psychopathic traits and autistic traits found in clinical populations is also found in a non-clinical population. This will be assessed by three self report questionnaires and one behavioural task (as described in 'Outcome Measures'). This investigation will also assess the potential link between of all of the traits measured and a specific SNP on the Oxytocin Receptor Gene (OXTR rs53576) to establish whether this mutation is associated with any of these behaviours.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at time of participation
* Proficient English reading comprehension

Exclusion Criteria:

* Current or previous diagnosis of a psychopathy, autism or related conditions.
* Not proficient in English reading comprehension

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is intended to be representative of the general population. Participants must be over 18 years of age, proficient in English comprehension and no current or previous diagnosis of psychopathy, autism or related conditions. Recruitment will not be excluded based on on ethnicity, nationality, sex, gender, religion, sexual orientation or any other characteristic.
  For the analysis of the behavioural traits investigated, 128 participants (58 male, 70 female) between the ages of 19 and 68 years (median age = 26) were included in the final analysis. For the genetic aspect of the study, 96 participants (40 male, 56 female) between the ages of 19 and 68 years (median age = 26) were included in the final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
31-item Questionnaire for Cognitive and Affective Empathy (QCAE) | 20 minutes
  Self-reported empathy levels. 19 items assessing cognitive empathy, 12 items assessing affective empathy. All items are rated on a Likert scale of agreement from 1 (strongly disagree) to 4 (strongly agree) with 4 items being reverse scored prior to analysis.
36-item 'Reading the Mind in the Eyes' behavioural task (RMET) | 20 minutes
  A behavioural task to assess a sub-scale of cognitive empathy, emotion recognition. RMET establishes an individual's ability to recognise the emotional state of strangers in photographs with only their eyes as visual cues, with each item consisting of a photograph of a stranger expressing a specific emotional state. Each item is scored as 1 for correct and 0 for incorrect, with a higher total score indicating a greater ability at recognising the emotional state of others.
26-item Levenson's Self-Report for Psychopathy (LSRP) | 20 minutes
  A self reporting questionnaire assessing psychopathic traits without the requirement fo a clinical assessment. 16 items assess primary psychopathy and 10 items assess secondary psychopathy. All items are rated on a Likert scale of agreement of 1 (strongly agree) to 4 (strongly disagree) with 7 items having their score reversed prior to analysis.
50-item Autism Quotient (AQ) | 20 minutes
  A self reporting questionnaire to assess autistic traits. The scale consists of 50 items, with 10 items fort each of the 5 subscales; social skill, attention switching, attention to detail, communication and imagination. Items are rated on a Likert scale of agreement from 0 (strongly or slightly disagree) to 1 (strongly or slightly agree), with 50% of the items being reversed prior to analysis.
OXTR rs53576 genotype | 3 days
  Saliva is collected from participants via passive drool, and stabiliser provided by the DNA extraction kit manufacturer is added (SalivaGene Collection Module II; Stratec Molecular GmbH). An extraction protocol provided by the kit manufacturer is followed to extract DNA from each saliva sample (PSP® SalivaGene 17 DNA Kit 1011, Stratec Molecular GmbH). Genotyping was carried out using a StepOnePlus thermocycler (Applied Biosystems) with a predesigned TaqMan® SNP genotyping assay for rs53576 with code C__3290335_10. Each DNA sample was run in duplicate and the PCR procedure was performed following manufacturer guidelines. Results will be flagged as either AA, AG or GG genotype.

CONTACTS AND LOCATIONS:
Overall Officials: Yiannis Mavrommatis, PhD, Principal Investigator — St. Mary's University, Twickenham; Kate Lawrence, PhD, Principal Investigator — St Marys University
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol — https://www.stmarys.ac.uk/staff-directory/jonathan-nixon